CLINICAL TRIAL: NCT07213778
Title: A Phase 3, Multicenter, Double-Blinded, Randomized Study to Evaluate REGN7508, a Factor XI Monoclonal Antibody, Versus Acetylsalicylic Acid for Prophylaxis of Symptomatic Venous Thromboembolism After Elective Total Knee Arthroplasty (ROXI-ASPEN)
Brief Title: REGN7508 Versus Acetylsalicylic Acid (ASA) for Venous Thromboprophylaxis After Total Knee Arthroplasty in Adult Participants
Acronym: ROXI-ASPEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R7508-DVT-24120; 2025-520479-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-03; First posted 2025-10-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Symptomatic Venous Thromboembolism (VTE)
Keywords: Total Knee Arthroplasty (TKA); Elective Unilateral TKA; Deep Vein Thrombosis (DVT); Pulmonary Embolism (PE)
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN7508 and Placebo (Experimental)
  Interventions: Drug: REGN7508; Drug: Placebo
- Placebo and ASA (Active Comparator)
  Interventions: Drug: Acetylsalicylic Acid (ASA); Drug: Placebo

INTERVENTIONS:
Drug: REGN7508 — Administered per the protocol
  Arms: REGN7508 and Placebo
Drug: Acetylsalicylic Acid (ASA) — Administered per the protocol
  Arms: Placebo and ASA
Drug: Placebo — Administered per the protocol

SUMMARY:
This study is researching an experimental drug called REGN7508 versus Acetylsalicylic Acid (ASA) (each called "study drug"). The study is focused on adults undergoing elective, unilateral (one side) total knee replacement surgery.

The aim of the study is to see how effective the study drug is at preventing Venous Thromboembolism (VTE) and other related diseases after total knee replacement surgery compared to acetylsalicylic acid.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Is undergoing a primary elective unilateral TKA
2. Is in good health based on laboratory safety testing as described in the protocol

Key Exclusion Criteria:

1. Any condition that, as assessed by the investigator, may confound the results of the study or pose an additional risk to the participant by study participation
2. History of bleeding in the 6 months prior to randomization requiring hospitalization or transfusion; history of intracranial or intraocular bleeding, excessive operative or post-operative bleeding, and traumatic spinal or epidural anesthesia; history of bleeding diathesis (eg, hemophilia A or B, von Willebrand's Factor deficiency)
3. History of thromboembolic disease or thrombophilia
4. History of platelet dysfunction
5. Has received or plans to receive preoperative enoxaparin on the day prior to TKA surgery

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite endpoint of symptomatic VTE and VTE-related death | Through day 30 visit

SECONDARY OUTCOMES:
Incidence of confirmed symptomatic Deep Vein Thrombosis (DVT) | Through day 30 visit
Incidence of confirmed Pulmonary Embolism (PE) | Through day 30 visit
Incidence of VTE-related death | Through day 30 visit
Time to first event of the composite endpoint of symptomatic VTE and VTE-related death | Through day 30 visit
Time to first event of confirmed symptomatic DVT | Through day 30 visit
Time to first event of confirmed PE | Through day 30 visit
Time to VTE-related death | Through day 30 visit
Incidence of the composite endpoint of major bleeding and Clinically Relevant Non-Major (CRNM) bleeding | Through day 30 visit
Incidence of minor bleeding | Through day 30 visit
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Through day 90 visit
Severity of TEAEs | Through day 90 visit
Incidence of Anti-drug Antibody (ADA) to REGN7508 | Through day 90 visit
Magnitude of ADA to REGN7508 | Through day 90 visit
Concentrations of REGN7508 | Through day 90 visit

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (9):
- United States (9):
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Medical Research of Westchester - MPLUS Research Network, Miami, Florida
  - Phoenix Clinical Research, Tamarac, Florida
  - NextStage Clinical Research, St. Francis Medical Park, Wichita, Kansas
  - Sinai Hospital of Baltimore, Inc., Baltimore, Maryland
  - Ohio Clinical Trials, Columbus, Ohio
  - HD Research - Memorial Hermann Village, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Spokane Joint Replacement Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/